CLINICAL TRIAL: NCT05391373
Title: Effect of Laughter Therapy on Perceived Stress and Quality of Life in Women With Breast Cancer: An Assessor-blinded, Parallel Group, Randomized Controlled Trial
Brief Title: Effect of Laughter Therapy on Perceived Stress and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Pinar Zorba Bahceli, PhD RN, Asistant Professor, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/271
Record Dates: First submitted 2022-05-21; First posted 2022-05-25 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Laughter Therapy
Keywords: Perceived stress; Quality of life; Laughter therapy; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter Therapy Group (Experimental): The women with breast cancer in the intervention group received two sessions of laughter therapy per week for eight weeks.Each laughter therapy session lasted 40 minutes.
  Interventions: Behavioral: Laughter therapy
- Control group (No Intervention): The control group did not receive any intervention during the study period.

INTERVENTIONS:
Behavioral: Laughter therapy — Each session started with a 10-minute breathing exercise accompanied by relaxing music, followed by 20-minute laughing exercises. Afterwards, the session was ended with a 10-minute meditation accompanied by relaxing music.
  Arms: Laughter Therapy Group

SUMMARY:
Breast cancer is the most common type of cancer seen in women worldwide and ranks first. Chemotherapy is one of the commonly used methods of treatment in breast cancer. Physiological and psychological symptoms that occur due to chemotherapy treatment affect women negatively and reduce their quality of life. For this reason, there is a need for an intervention that could decrease psychological symptoms such as stress and improve quality of life in women with breast cancer. In the literature, it is stated that laughter therapy which is one of the non-pharmacological methods, can be an effective nursing intervention to decrease stress and improve the quality of life in women with breast cancer.

DETAILED DESCRIPTION:
This an assessor-blinded, parallel group randomized controlled trial aimed that investigating the effect of laughter therapy on perceived stress and quality of life in women with breast cancer.This trial was conducted in the chemotherapy outpatient clinic of training and research hospital located in Turkey. All patients were women with breast cancer who received a once-weekly Paclitaxel regimen.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older women,
* Stages II or III breast cancer
* Receiving Pacitaxel chemotherapy regimen per a week

Exclusion Criteria:

* Using any complementary and alternative (CAM) treatment method during practice
* Having psychological diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-12 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | The scale was filled in the baseline (before the beginning of the Laughter therapy), 5th and 9th weeks.
  The scale consists of 14 items in total and was designed to measure how stressful the changing situations in the individual's life are perceived.The scale is a 5-point Likert-type scale with each item ranging from "never (0)" to "very often (4)". 7 of the scale items with positive expressions are scored in reverse and the total score that can be obtained from the scale ranges from 0 to 56. Eskin et al. performed the validity and reliability study of the Turkish version of Perceived Stress Scale and the internal consistency of the scale was determined to be 0.82.

SECONDARY OUTCOMES:
Quality of Life Scale (SF-12) | The scale was filled in the baseline (before the beginning of the Laughter therapy), 5th and 9th weeks.
  The scale evaluates the quality of life of individuals.The scale consists of 12 items and two sub-dimensions in total.While the items related to physical and emotional role were answered as yes or no, the other items had likert type options ranging between 3 and 6. While the Physical Component Summary-12 (PCS-12) score was obtained from the sub-dimensions of general health, physical functionality, physical role and body pain; The Mental Component Summary-12 (MCS-12) score was obtained from the sub-dimensions of social functionality, emotional role, mental health and energy. Both the PCS-12 and MCS-12 scores range from 0 to 100, with the higher score representing better health.Soylu et al. performed the validity and reliability study of the Turkish version of Quality of Life Scale (SF-12) and the internal consistency of the scale was determined to be 0.73.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Bakircay University Health Sciences Faculty, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No